CLINICAL TRIAL: NCT03668314
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of Single and Multiple Doses of Orally Administered RDN-929 in Healthy Adult and Elderly Subjects
Brief Title: Single and Multiple Ascending Dose and Food Effect PK Study in Healthy Adult and Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Collaborators: QPS Netherlands B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RDN-929-101
Record Dates: First submitted 2018-09-06; First posted 2018-09-12 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Parts 1 and 3 are parallel designs with escalating doses within each part. Part 2 is a FE cross-over study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1:1 - 1:6 RDN-929 (Experimental): RDN-929 single dose capsule
  Interventions: Drug: RDN-929
- Cohort 1:1 - 1:6 placebo (Placebo Comparator): Placebo single dose capsule
  Interventions: Drug: Placebo oral capsule
- Cohort 2:1 (Experimental): Fed/Fast RDN-929
  Interventions: Drug: RDN-929 TBD dose
- Cohort 3:1- 3:4 RDN-929 (Experimental): RDN-929 multiple dose capsules once daily for 12 days
  Interventions: Drug: RDN-929
- Cohort 3:1- 3:4 placebo (Placebo Comparator): placebo multiple dose capsules once daily for 10 days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: RDN-929 — Single dose from 2 mg to TBD
  Arms: Cohort 1:1 - 1:6 RDN-929
Drug: Placebo oral capsule — Matching placebo Single dose
  Arms: Cohort 1:1 - 1:6 placebo
Drug: RDN-929 TBD dose — Fed vs fast dose TBD based upon results of previous cohorts
  Arms: Cohort 2:1
Drug: RDN-929 — Multiple dose based on results of previous cohorts
  Arms: Cohort 3:1- 3:4 RDN-929
Drug: Placebo oral capsule — Matching placebo multiple dose
  Arms: Cohort 3:1- 3:4 placebo

SUMMARY:
A three (3) part study to evaluate the safety, tolerability and PK of RDN-929

DETAILED DESCRIPTION:
Part 1 (Randomized, Double Blind):

Up to 6 single ascending doses of RDN-929 are planned to be tested in 6 cohorts of 8 healthy males (Cohort 1:1 to 1:6). Within each cohort subjects will be randomly assigned to receive either a single dose of RDN-929 (6 subjects) or matched placebo (2 subjects).

Part 2 (Open):

Part 2 will consist of 2 crossover treatment periods in one cohort of 12 healthy elderly subjects (at least 3 of each gender), aged 55-80 years. The treatments will be separated by a washout period of at least 7 days. The dose selected for this part of the study will be based on the results of Part 1.

In Period 1, subjects will be randomized to receive a single dose of RDN-929 in either fasted or fed status. In Period 2, subjects will receive a single dose of RDN-929 under the alternate status.

Part 3 (Randomized, Double Blind):

Multiple ascending doses (MAD) of RDN-929 are planned to be tested in up to 4 cohorts of 8 healthy elderly subjects (at least 3 of each gender per dose level cohort), aged 55-80 years. The doses will be selected by the safety review committee (SRC) based on all available safety, tolerability and PK data and after approval by the ethics committee.

Within each cohort subjects will be randomly assigned to receive either, RDN-929 once daily (6 subjects) or matched placebo (2 subjects) once daily for 12 days. Escalation to the next higher dose level will be based upon a review of the safety and tolerability data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the Investigator, based on a medical evaluation including medical history physical examination, neurological examination, laboratory tests and cardiac monitoring
* Men, age 18-54 years inclusive at Screening (Part 1) or men and postmenopausal or surgically sterile women age 55-80

Exclusion Criteria:

* Any history of major psychiatric disorders, including substance use disorders, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria.
* Acute suicidality or history of suicidal behavior.
* Alanine aminotransferase or aspartate aminotransferase levels greater than 1.5 times the upper limit of normal (ULN) at Screening. One retest is allowed.
* A corrected QT interval measurement corrected according to the Fridericia rule (QTcF) > 450 msec during controlled rest at screening or between screening and first dose administration, or family history of long QT syndrome.
* Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, in the judgement of the Investigator or Medical Monitor, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
* A clinically significant vital signs abnormality at screening or between screening and first dose administration. This includes, but is not limited to, the following, in the supine position: (a) systolic blood pressure < 90 or >150 mmHg, (b) diastolic blood pressure <50 or > 95 mmHg, or (c) heart rate < 45 or >100 beats per minute.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Screening to end of study, up to 7 weeks
  Listing and summary of AE incidence
Number of subjects with Physical exam findings | Screening to end of study, up to 7 weeks
  Listing of clinically significant changes in PE findings
Number of subjects with Clinical safety lab changes | Screening to end of study, up to 7 weeks
  Listing and change from baseline to end of study
Number of subjects with Systolic blood pressure changes | Screening to end of study, up to 7 weeks
  Listing and change from baseline to end of study
Number of subjects with Heart rate changes | Screening to end of study, up to 7 weeks
  Listing and change from baseline to end of study
Number of subjects with 12 Lead ECG changes | Screening to end of study, up to 7 weeks
  Change in 12-lead ECG parameters from baseline to end of study
Number of subjects with 3 Lead ECG findings | Predose to 8 hours post dose on Day 1 (Parts 1 and 2) and Days 1 and 12 (Part 3)
  Listing of findings
Number of subjects with C-SSRS changes | Baseline to end of study (Part 3 only), up to 7 weeks
  Listing of results
Number of subjects with Visual analogue scale changes | Baseline to end of study for Part 1 and 3, up to 7 weeks
  VAS for headache and nausea

SECONDARY OUTCOMES:
Maximum observed plasma concentration, Cmax | Predose to 48 hours post first and last dose, up to 2 days (Parts 1 and 2) and 2 weeks (Part 3)
  Of RDN-929 and primary metabolite
Time to reach maximum observed plasma concentration, Tmax | Predose to 48 hours post first and last dose, up to 2 days (Parts 1 and 2) and 2 weeks (Part 3)
  Of RDN-929 and primary metabolite
Area Under the plasma concentration time curve, AUC | Predose to 48 hours post last dose, up to 2 days (Parts 1 and 2) and 2 weeks (Part 3)
  Of RDN-929 and primary metabolite

CONTACTS AND LOCATIONS:
Overall Officials: PI, Principal Investigator — QPS Holdings LLC
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands